CLINICAL TRIAL: NCT05056220
Title: A Randomized Multicentre, Double-Blinded and Placebo-Controlled, Trial of Human Albumin in the Treatment of Decompensated Cirrhosis Guided by the MICROB-PREDICT Biomarker
Brief Title: Personalized Long-term Human Albumin Treatment in Patients With Decompensated Cirrhosis and Ascites
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aleksander Krag (Other)
Collaborators: EASL - CLIF Consortium (Other)
Responsible Party: Sponsor-Investigator, Aleksander Krag, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-501006-34-01; 825694 (Other Grant/Funding Number: HORIZON 2020)
Record Dates: First submitted 2021-09-20; First posted 2021-09-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Decompensated Cirrhosis and Ascites
MeSH Terms: conditions — Ascites | interventions — Serum Albumin, Human; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: There will exist two levels of masking in the current trial. Masking of biostratification outcome (high expected effect of human albumin or low expected effect of human albumin): Participant, Investigator and Outcome Assessor Masking of treatment assignment (human albumin 20% or saline 0.9%): Participant and Outcome Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High expected effect: Human Albumin 20% + Standard Medical Treatment (Active Comparator): Participants stratified to a high expected effect of human albumin and randomized to active treatment with 20% Human Albumin infusions.
  Interventions: Drug: Human albumin
- High expected effect: Saline (NaCl 0.9%) + Standard Medical Treatment (Placebo Comparator): Participants stratified to a high expected effect of human albumin and randomized to placebo treatment with 0.9% NaCl (saline) infusions.
  Interventions: Drug: sodium chloride
- Low expected effect: Human Albumin 20% + Standard Medical Treatment (Active Comparator): Participants stratified to a low expected effect of human albumin and randomized to active treatment with 20% Human Albumin infusions.
  Interventions: Drug: Human albumin
- Low expected effect: Saline (NaCl 0.9%) + Standard Medical Treatment (Placebo Comparator): Participants stratified to a low expected effect of human albumin and randomized to placebo treatment with 0.9% NaCl (saline) infusions.
  Interventions: Drug: sodium chloride

INTERVENTIONS:
Drug: Human albumin — 20% Human Albumin infusions (every 10th day +/- 4 days) with dosing according to the participants bodyweight (1.5 grams of albumin per kg bodyweight with a maximum of 100 grams)
  Arms: High expected effect: Human Albumin 20% + Standard Medical Treatment; Low expected effect: Human Albumin 20% + Standard Medical Treatment
Drug: sodium chloride — 0.9% NaCl infusions (every 10th day +/- 4 days) with dosing according to the corresponding volume used of 20% Human Albumin (1.5 grams of albumin per kg bodyweight with a maximum of 100 grams)
  Arms: High expected effect: Saline (NaCl 0.9%) + Standard Medical Treatment; Low expected effect: Saline (NaCl 0.9%) + Standard Medical Treatment

SUMMARY:
The goal of this clinical biomarker validation trial is to test the effect of a predictive biomarker panel to human albumin infusions in patients with liver cirrhosis and ascites. The main questions it aims to answer are:

* If the predictive biomarker panel can identify patients who are likely to benefit from regular human albumin infusions
* If the predictive biomarker panel can lower the number-needed-to-treat of regular human albumin infusions in patients with liver cirrhosis and ascites

The predictive biomarker panel will stratify patients into either a high- or low-expected effect of human albumin infusions. Hereafter are participants randomized into treatment arms.

Participants in the active treatment arm will receive regular human albumin infusions during a course of 6 months. Infusions will occur every 10th day for the duration of the study.

Researchers will compare 20% human albumin infusions with regular 0.9% sodium chloride to identify the effects on the number of liver-related events.

ELIGIBILITY:
Inclusion Criteria:

* Decompensated liver cirrhosis defined as Child-Pugh score 7-12
* Clinical and/or ultrasound evidenced ascites
* Age ≥ 18 years
* At least five days since resolution of a decompensation event or any condition requiring hospitalisation

Exclusion Criteria:

* Patients with acute or subacute liver failure without underlying cirrhosis
* Patients with cirrhosis who develop decompensation in the postoperative period following partial hepatectomy
* Refractory ascites as defined by the International Ascites Club
* Existing TIPS inserted <6 months ago
* Portal vein thrombosis without signs of cavernous transformation or recanalization
* Severe alcoholic hepatitis (Glasgow Alcoholic Hepatitis Score > 11)
* Hepatic encephalopathy grade III-IV
* Current, planned or previous treatment with direct antiviral agents for hepatitis C virus (HCV) in the last six months Contraindications for human albumin infusion (pulmonary oedema, hypersensitivity etc.)
* Evidence of current malignancy except for non-melanocytic skin cancer and hepatocellular carcinoma within Barcelona Clinic Liver Cancer (BCLC)-0 or BCLC-A
* Presence or history of severe extra-hepatic diseases (e.g.,chronic renal failure requiring hemodialysis, severe heart disease (NYHA > II); severe chronic pulmonary disease (GOLD Score ≥ C), severe neurological and psychiatric disorders, pulmonary arterial hypertension)
* HIV positive or other condition associated with and/or requiring immunosuppression
* Previous liver or other transplantation
* Pregnancy
* Breastfeeding
* Patients who decline to participate, patients who cannot provide prior written informed consent due to other causes than hepatic encephalopathy or patients with hepatic encephalopathy who cannot provide prior written informed consent and when there is documented evidence that the patient has no legal surrogate decision maker or sufficient ability to provide delayed informed consent
* Physician's denial (investigator considers that the patient will not adhere to the study protocol scheduled, e.g. in case of heavy drinking)
* Participation in another study within 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Cumulative number of liver-related clinical outcomes | 6 months
  Cumulative number of liver-related clinical outcomes (variceal bleeding, ascites, spontaneous bacterial peritonitis, infection requiring hospitalization, acute kidney injury and overt hepatic encephalopathy) and TIPS (insertion or revision) with death and liver transplantation as counting and censoring events

SECONDARY OUTCOMES:
6-months survival | 6 months
The number of episodes of acute-on-chronic liver failures | 6 months
  Acute-on-chronic liver failure (ACLF) is defined according to the CLIF-C ACLF definition.
Number of organ failures | 6 months
  Where an organ failure is defined according to the CLIF-C ACLF definition.
Time-to-first liver-related clinical outcome | 6 months
  A liver-related clinical outcome is defined as variceal bleeding, ascites, spontaneous bacterial peritonitis, infection requiring hospitalization, acute kidney injury (>=1B), overt hepatic encephalopathy, TIPS insertion, liver transplantation or death. Time to any of these outcomes are defined as the time from trial inclusion until 1) the date of diagnosis of any of the complications, 2) the date of the procedure (TIPS or liver transplantation) or date of death.
Change in SF-36 | 6 months
  Quality of life for participants, as measured by Short Form 36 (SF-36), ranging from 0 to 100 with a score of 0 equal to maximum disability and score of 100 no disability.
Change in CLDQ | 6 months
  Quality of life for participants, as measured by the Chronic Liver Disease Questionnaire (CLDQ), consisting of 29 items within 7 domains. Response on a Likert scale ranging from 1 (most impairment) to 7 (least impairment). Total score by adding score for each item and divide by number of items (29).
Change in EQ-5D-5L | 6 months
  Quality of life for participants, as measured by the EuroQoL-5 Domain, 5 levels (EQ-5D-5L). Consist of 5 domains with 5 levels where the lowest level (1) is the worst imaginable health and highest level (5) is the best imaginable health.
Time to first hospital admission (in days) | 180 days
Number of hospital admissions | 180 days
Days spent on hospitalization (in days) | 180 days
Number of intensive care unit admissions | 180 days
Length of intensive care unit admissions (in days) | 180 days
Number of large volume paracentesis | 6 months
Analysis of the cost/effectiveness ratio | 6 months
  Analyzed by an incremental cost-effectiveness ratio (ICER) calculation
Health economic evaluation | 6 months
  Analyzed by the change in quality-adjusted life years (QALYs) relative to the ICER.
Changes in serum albumin levels | 6 months
  Measured from baseline and throughout the trial in grams per litre (g/L)
Number of treatment-related adverse events | 6 months
  Adverse events which are deemed related to the trial intervention
Number of treatment-related serious adverse events | 6 months
  Adverse events which are deemed related to the trial intervention
Signatures associated with a poor prognosis as defined by the Microb-Predict biomarker | 6 months
  Change in concentration of the panel of predictive circulating metabolites compared to metabolite levels in other body fluid compartments (blood, urin, stool and saliva)
Incidence of refractory ascites | 6 months
Incidence of variceal bleeding | 6 months
Incidence of spontaneous bacterial peritonitis | 6 months
Incidence of infection requiring hospitalization | 6 months
Incidence of acute kidney injury >= 1B | 6 months
  According to the Kidney Disease: Improving Global Outcomes (KDIGO) definition ranging from stage 1A to 3 where a higher stage is worse.
Incidence of hepatorenal syndrome acute kidney injury | 6 months
Incidence of overt hepatic encephalopathy | 6 months
Incidence of liver transplantation | 6 months
Incidence of TIPS insertion or revision | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Aleksander Krag, Professor, Principal Investigator — Odense University Hospital
Locations (12):
- Katholieke Universiteit Leuven, Leuven, Belgium
- Denmark (2):
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Münster, Münster
- Debreceni Egyetem, Debrecen, Hungary
- Netherlands (2):
  - Academisch Ziekenhuis Leiden, Leiden
  - Alrijne Ziekenhuis Leiden, Leiderdorp
- Spain (2):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Del Mar, Barcelona
- King's College Hospital, London, United Kingdom

REFERENCES:
- [Derived] Torp N, Israelsen M, Coenraad M, Papp M, Shawcross D, Korenjak M, Angeli P, Laleman W, Juanola A, Gines P, Trebicka J, Krag A; MICROB-PREDICT Consortium. Personalised human albumin in patients with cirrhosis and ascites: design and rationale for the ALB-TRIAL - a randomised clinical biomarker validation trial. BMJ Open. 2024 Feb 14;14(2):e079309. doi: 10.1136/bmjopen-2023-079309. PMID 38355195